CLINICAL TRIAL: NCT03776929
Title: Dialectical Behavioral Therapy in High Risk OrthopaedicTrauma Patients
Acronym: OI-DBT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is temporarily suspended until resources are put in place for enrollment
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Ida Leah Gitajn, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D18154
Record Dates: First submitted 2018-11-15; First posted 2018-12-17 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Fracture; Surgery
Keywords: Dialectical Behavioral Therapy; Orthopaedic; Trauma; Pain Catastrophizing Scale
MeSH Terms: conditions — Fractures, Bone; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): No intervention - Standard care only. Group of 32 subjects
- Dialectical Behavioral Therapy (Experimental): Dialectical Behavioral Therapy in addition to standard care. Four hour and a half group sessions (or one-on-one sessions, if not enough for a group session) commencing after surgery while still inpatient. Each session is designed to stand-alone, allowing for enrolling patients on a rolling basis.
  Interventions: Behavioral: Dialectical Behavioral Therapy

INTERVENTIONS:
Behavioral: Dialectical Behavioral Therapy — Dialectical Behavior Therapy (DBT) is a cognitive behavioral therapy that focuses on the balance between change and acceptance. DBT skills include four modules: two that enforce acceptance-oriented skills, mindfulness and distress tolerance, and two that promote change-oriented skills, interpersonal effectiveness and emotional regulation.
  Arms: Dialectical Behavioral Therapy

SUMMARY:
Psychological factors can affect the experience of pain and functional recovery from orthopedic injury. The purpose of this study is to examine the effect of brief Dialectical Behavior Therapy (DBT), a form of psychotherapy, on changing thoughts, feelings, and behaviors that can cause problems in daily living and interfere with recovery from orthopedic injury in patients who are at high risk for chronic pain and disability.

DETAILED DESCRIPTION:
Musculoskeletal injuries represent one of the leading causes of hospital admissions for adults, and often results in long term pain, poor function, and permanent disability. Patients afflicted with musculoskeletal injuries contribute to an enormous cost to society in terms of direct health care spending, as well as indirect costs related to permanent disability, loss of work, and chronic pain contributing to the rising opioid epidemic. This is clearly a substantial and costly issue at Dartmouth-Hitchcock Medical Center (DHMC) as well as the country at large. From 2011 to 2017, 54% of patients who were admitted for fracture at DHMC had either a psychiatric diagnosis and/or a substance abuse diagnosis. It is likely that this number vastly underestimates the true amount of emotional distress present in this patient population because many patients with these issues do not carry formal psychiatric diagnoses. Diagnosis of psychiatric illness or substance abuse was associated with significantly higher resource utilization during hospital admission in terms of hospital length of stay (LOS, mean difference 3 days), need for ICU stay, number of consulting services, disposition to rehab, and rate of unplanned readmissions (21% versus 39%, respectively). Furthermore, this patient population had significantly higher mean pain score during admission and required 10-fold more opioids prescribed [measured in total morphine equivalents (MME)] and number of separate prescriptions needed.

These data within the investigator's own patient population reinforce the well documented reciprocal association between chronic pain and adverse mental health outcomes, such that pain triggers depression for example, but depression may as well exacerbate experiences of pain. In fact, catastrophic thinking about pain (tendency to assume the worst and believe that one will be unable to cope with the outcome), pain anxiety, and symptoms of depression are key factors that explain the magnitude of disability and pain intensity after musculoskeletal trauma. Resilience, the capacity to adapt to or recover from adversity, has been shown to attenuate the association between depression and pain. For this reason, the investigators believe it is important for patients to learn effective coping skills in order to effectively manage their pain and fear associated with recovering from a traumatic injury.

Dialectical Behavior Therapy (DBT) is a cognitive behavioral therapy that focuses on the balance between change and acceptance. DBT skills include four modules: two that enforce acceptance-oriented skills, mindfulness and distress tolerance, and two that promote change-oriented skills, interpersonal effectiveness and emotional regulation. This psychosocial treatment aims to reduce ineffective action tendencies associated with dysregulated emotions. DBT has been studied extensively in adult samples, across a wide range of settings. It has been shown to be effective in management of intense emotional states and development of coping skills in the most challenging patient populations including patients with Borderline Personality Disorder (BPD), eating disorders, and substance abuse. Furthermore, DBT-based interventions have demonstrated preliminary effectiveness in managing chronic pain and pain catastrophizing and anxiety. As such, patients with orthopedic trauma at high risk for chronic pain and disability would benefit from an evidence-based treatment approach that would teach them how to change thoughts, feelings, and behaviors that could cause problems in daily living and interfere with recovery from injury.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Admitted to Dartmouth-Hitchcock Medical Center with an operatively treated fracture.

Exclusion Criteria:

* Non-English speaking
* Pain Catastrophizing Scale (PCS) score of < 13
* Anticipating hospital length of stay of less than 2 days
* Are expected to have severe problems maintaining follow-up and treatment recommendations
* Have current or impending incarceration
* Are actively psychotic or manic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change over time in Pain Severity: VAS | Baseline, 2 week follow-up, 6-8 week follow-up, 10-14 week follow-up
  Visual Analogue Scale (VAS) Pain scores documented in the patient's medical record. Score Range 0-10. Higher score indicates greater pain.
Number of Opioids Administered | Hospital admission to hospital discharge, approximately 4-7 days
  The opioids administered during hospitalization measured in total morphine equivalents

SECONDARY OUTCOMES:
Change over time in General Health Status | Baseline, 2 week follow-up, 6-8 week follow-up, 10-14 week follow-up
  Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health: 10-item measure of physical and mental health. Scale range 0 to 100, mean 50, standard deviation 10. A higher score represents a better outcome.
Change over time in Psychological Functioning - Depression | Baseline, 2 week follow-up, 6-8 week follow-up, 10-14 week follow-up
  Patient Health Questionnaire-9 (PHQ-9): 9-item measure of major depression symptom severity on a 4-point Likert-type scale. Score range 0-27; Higher score indicates more severe depressive symptoms.
Change over time in Psychological Functioning - PTSD | Baseline, 2 week follow-up, 6-8 week follow-up, 10-14 week follow-up
  PTSD Checklist for DSM-5 (PCL-5): 20-item measure of DSM-5 PTSD symptom severity on a 5-point Likert-type scale. Scale range 0-80. Higher score indicates more severe PTSD symptoms
Change over time in Pain Anxiety: PASS-20 | Baseline, 2 week follow-up, 6-8 week follow-up, 10-14 week follow-up
  Pain Anxiety Symptoms Scale (PASS-20): 20-item measure of pain anxiety on a 6-point Likert-type scale. Scale range 0-100. Higher score indicates more pain-related anxiety
Change over time in Pain Interference: BPI-SF | Baseline, 2 week follow-up, 6-8 week follow-up, 10-14 week follow-up
  Brief Pain Inventory-Short Form (BPI-SF): 9-item measure of pain severity and impact of pain on daily functions. This is a 10-point scale with 0 being the best possible score, meaning "no pain", and 10 being the worst possible score, meaning "pain as bad as you can imagine".

CONTACTS AND LOCATIONS:
Overall Officials: Ida L Gitajn, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock, Lebanon, New Hampshire, United States